CLINICAL TRIAL: NCT00289302
Title: InSync Implantable Cardioverter Defibrillator Registry: Cardiac Resynchronization Therapy
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Other Study IDs: 196
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2006-09

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: Heart Failure; Cardiac pacing; Cardiac resynchronization therapy; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: Cardiac resynchronization therapy device

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy (CRT) may be prescribed. CRT is similar to a pacemaker. It is placed (implanted) under the skin of the upper chest. CRT is delivered as tiny electrical pulses to the right and left ventricles through three or four leads (soft insulated wires) that are inserted through the veins to the heart.

People who have a dangerously fast heart beat, or whose heart is at risk of stopping beating, may be in need of an electronic device called an implantable cardioverter defibrillator (ICD). An ICD is implanted surgically just under the skin in the upper chest area and it sends a strong electrical impulse, or shock, to the heart to return it to a normal rhythm. If the heart is beating too slowly or at an abnormal rhythm, an ICD can also pace the heart to return the heart to its normal rhythm. The InSync ICD device can change the timing of when the left and right ventricles of the heart are paced to beat.

The purpose of this study is to monitor the long-term performance of the InSync ICD Model 7272 and the InSync Marquis 7277 systems for cardiac resynchronization therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with the InSync ICD or InSync Marquis cardiac resynchronization therapy (CRT) system (includes InSync ICD Model 7272 or InSync Marquis Model 7277, right atrial lead, right ventricular lead and any market released Medtronic left ventricular lead or the investigational Attain Model 4189 lead which was implanted during the MIRACLE ICD Study)

Exclusion Criteria:

* Patients with a history of a previously failed placement of a currently investigational Medtronic left ventricular lead within 30 days of enrollment in the InSync ICD Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: InSync ICD Registry Study Leader, Study Chair — Medtronic
Locations (51):
- United States (51):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - San Diego, California
  - Stanford, California
  - New Haven, Connecticut
  - Newark, Delaware
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Palm Beach Gardens, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Oak Lawn, Illinois
  - Indianapolis, Indiana
  - Davenport, Iowa
  - Des Moines, Iowa
  - Topeka, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Houma, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Cherry Hill, New Jersey
  - Hackensack, New Jersey
  - Albany, New York
  - Chapel Hill, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mayfield Heights, Ohio
  - Oklahoma City, Oklahoma
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Providence, Rhode Island
  - Spartanburg, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin